CLINICAL TRIAL: NCT06432985
Title: Contingency Management for Veteran Smokers With or at Risk for Cancer
Brief Title: Smoking Cessation CM for Veterans With or at Risk for Cancer
Acronym: CM_TUD_Cancer
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Collaborators: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NURA-006-23F; 24-40951 (Other: University Of California, San Francisco)
Record Dates: First submitted 2024-05-20; First posted 2024-05-29 (Actual); Last update posted 2025-09-30 (Actual); Status verified 2025-09

CONDITIONS: Tobacco Use Disorder; Substance Use Disorder
Keywords: Tobacco; Contingency Management; Lung Cancer
MeSH Terms: conditions — Tobacco Use Disorder; Substance-Related Disorders; Lung Neoplasms | interventions — Focus Groups; Behavior Therapy; Cognitive Behavioral Therapy

STUDY DESIGN:
Intervention Model Description: Parallel Assignment
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Focus Group (Other): The investigators will iteratively develop an acceptable mobile CM protocol using qualitative feedback from Veterans in VA patients in LCS or in cancer care and LCS and oncology staff.
  Interventions: Behavioral: Focus Group
- Contingency Management (Experimental): Veterans in VA LCS or cancer care will receive mobile CM plus behavioral counseling and cessation medication over 5 weeks.
  Interventions: Behavioral: Contingency Management; Behavioral: Behavioral Counseling (Cognitive Behavioral Therapy, CBT)
- TUD Treatment as Usual (Active Comparator): Participants assigned to TAU will receive time-matched Medication Management plus usual care (referral to VA Tobacco Cessation Clinic and provision of the VA Telequit quitline).
  Interventions: Behavioral: Behavioral Counseling (Cognitive Behavioral Therapy, CBT); Behavioral: TUD Treatment as Usual (TAU)

INTERVENTIONS:
Behavioral: Focus Group — In 60-minute focus groups, participants will be categorized based on their survey responses and engaged in semi-structured discussions using open-ended questions and probes to gather detailed information. The moderators will follow best practices in qualitative research, introducing the topic of smoking cessation in the context of cancer screening and treatment and guiding the discussions from broader issues to participant-generated examples.
  Arms: Focus Group
Behavioral: Contingency Management — Participants will provide baseline data on their recent substance use and smoking habits and severity. They will receive a CO monitor and iCO app and will upload videos verifying smoking abstinence a minimum of once per day, 5 times per week. Financial incentives will be provided at weekly visits contingent on tobacco abstinence verified through Remote (mobile) CO monitoring. They will receive clinician feedback at the time of each CO reading, following established VA protocols for CM.
  Arms: Contingency Management
Behavioral: Behavioral Counseling (Cognitive Behavioral Therapy, CBT) — Participants will receive a 5-session smoking cessation behavioral counseling for approximately 15-20 minutes weekly. Sessions may be held by secure video conference or by telephone, per participant preference. Sessions will use CBT principles with MI incorporated for resolving reluctance to quit.
  Arms: Contingency Management; TUD Treatment as Usual
Behavioral: TUD Treatment as Usual (TAU) — Participants assigned to TAU will receive referral to VA Tobacco Cessation Clinic and provision of the VA Telequit quitline. The VA Tobacco Cessation Clinic is modeled after VA Tobacco Cessation Clinics across all VA facilities and involves delivery of brief counseling and pharmacotherapy for TUD if desired. VA Telequit is a national toll-free number available to Veterans that allows them to speak with a smoking cessation counselor for a recommended minimum of five sessions to develop a quit plan and receive counseling, strategies to prevent relapse, and weekly proactive follow-up calls based on National Cancer Institute guidelines.
  Arms: TUD Treatment as Usual

SUMMARY:
Tobacco use among US Veterans poses significant health problems and challenges to their overall well-being. The aim of this project is to evaluate the effectiveness of a program called Contingency Management (CM) in helping Veterans quit smoking during lung cancer screening or cancer care at VA clinics. CM is a behavioral treatment that uses rewards to encourage smoking cessation when verified through biological testing. In the first year, the researchers will develop a mobile CM protocol based on feedback from Veterans and healthcare staff through focus groups. In the second year, they will conduct a pilot study to test the feasibility of the mobile CM program along with counseling and medication for 20 Veterans over a five-week period. The success of the pilot study will determine whether to proceed with a larger randomized controlled trial (RCT) in years three to six, comparing the efficacy of mobile CM with standard treatment. The project will take place at SFVA.

DETAILED DESCRIPTION:
Smoking at the time of lung cancer screening (LCS) or cancer diagnosis is associated with treatment failure, shortened lifespan, and diminished quality of life. Beyond the increased morbidity and mortality, smoking after a cancer diagnosis is associated with an estimated $3.4 billion in healthcare costs. Despite these risks, the VA does not routinely integrate smoking cessation treatment into LCS screening or cancer care, and quit rates are low.

Contingency Management (C) is a behavioral therapy approach that reinforces desired behaviors, such as smoking cessation, through the provision of tangible rewards or incentives. The goal of this Proof of Concept and Clinical Trial project is to evaluate the acceptability, feasibility, and efficacy of Contingency Management (CM) for smoking cessation among Veterans in lung cancer screening (LCS) or cancer care in Veterans Affairs (VA) clinics.

Research indicates that CM must be tailored to the clinical population and context. This staged investigation will occur in three phases. First, the investigators will conduct Focus Groups, to iteratively develop an acceptable mobile CM protocol using qualitative feedback from Veterans in VA patients in LCS or in cancer care and LCS and oncology staff. Afterward, the investigators will conduct a Pilot Study to examine the feasibility of mobile smoking cessation CM with for VA patients in LCS or in cancer care. In a single arm study, Veterans in VA LCS or cancer care will receive mobile CM plus behavioral counseling and cessation medication over 5 weeks. If successful, the investigators will conduct a Randomized Controlled Trial (RCT) to assess efficacy of mobile CM compared with treatment as usual (TAU). Veterans diagnosed with cancer or in LCS will be randomized to receive a 5-week CM condition (CM plus behavioral counseling) or TAU (referral to VA Tobacco Cessation Clinic and VA quitline). Both groups will receive pharmacotherapy.

The primary aims of this study are to develop an acceptable mobile CM protocol through qualitative feedback from Veterans and VA staff, to examine the feasibility of mobile smoking cessation CM among Veterans in LCS or cancer care through a pilot study, and to assess the efficacy of mobile CM compared to treatment as usual through a randomized controlled trial among Veterans diagnosed with cancer or in LCS.

ELIGIBILITY:
Inclusion Criteria:

In order to be eligible to participate in this study, an individual must meet all of the following criteria:

* Human Subjects Involvement and Characteristics: This Proof of Concept and Clinical Trial has three stages. The Proof-of-Concept Phase (Years 1-2) includes a Focus Group phase (Year 1) in which the investigators will recruit both Veterans and non-Veterans (VA clinical staff); and a Pilot Study (Year 2) in which the investigators will recruit Veterans in LCS or cancer treatment at San Francisco VA Healthcare System (SFVAHCS). If the Pilot Study is successful, the investigators will recruit Veterans in LCS or cancer treatment for the RCT (Years 3-6).
* Focus Groups: For Focus Groups (Year 1), the investigators will recruit both Veterans and VA clinical staff at SFVAHCS.

Veterans:

* Age 18 years or older
* Veteran eligible for VA healthcare
* English-speaking
* Received SFVAHCS cancer monitoring or treatment or LCS within the past 24 months
* Active cigarette smoking within the past 24 months
* Have access to Wi-Fi and a device that supports audio and video communication

VA Clinical Staff:

* Current member of clinical staff at the SFVAHCS
* Have participated in the care of at least 5 VA cancer or LCS patients in the past 6 months

Pilot Feasibility Study (Year 2) and Randomized Controlled Trial

Inclusion criteria:

* Age 18 years or older
* Veteran currently receiving medical care at SFVAHCS (at least one clinical visit same calendar year for cancer)
* English-speaking
* Current, active (same calendar year) enrollment in VA LCS, or current (same calendar year) diagnosis of cancer documented in the VA medical record, confirmed through medical record review
* Current (past 30 days) cigarette smoking a minimum of 1 cigarette per day (average), assessed by Timeline Followback (TLFB)92, 99-101
* Open to receiving smoking cessation interventions

Exclusion Criteria:

Focus Groups: For Focus Groups (Year 1), the investigators will recruit both Veterans and VA clinical staff at SFVAHCS.

Veterans:

Exclusion criteria: Assessed by Co-PIs' medical record review:

* Current severe, untreated mental illness (i.e., psychosis, bipolar disorder, and/or substance use disorder (SUD)) and/or
* Current (past 30 days) active suicidal/homicidal ideation or severe behavioral instability that would prevent participation
* Never smokers or quit smoking for longer than 36 months prior to consent (4) no access to Wi-Fi or devices that support audio and video communication

VA Clinical Staff:

Exclusion Criteria:

* Unable to commit 1.5 hours (60 min focus group and self-report questionnaires)

Pilot Feasibility Study (Year 2) and Randomized Controlled Trial

Exclusion Criteria:

* An individual who meets any of the following criteria will be excluded from participation in this study:
* Evaluated by investigative team medical record review and clinical assessment:
* Psychotic disorders, bipolar disorder, neurocognitive disorder, substance use disorders, or other psychiatric or medical conditions judged by the PI to be unstable in the past 30 days, based on screening results and/or medical record review, including conditions for which large sums of money would be potentially destabilizing
* Untreated, current, active problem gambling, assessed by medical record diagnosis and/ or Problem Gambling Severity Index (PGSI) score 8
* Metastatic cancer or enrollment in end of life/ palliative care
* Unable to commit to time commitment required for participation
* Currently pregnant or planning to become pregnant during the study (people of childbearing potential ages 18-55 who are pregnant or state that they plan to become pregnant during the study)
* A suicide attempt or suicidal ideation with intent in the 30 days prior to enrollment
* Concurrent enrollment in a tobacco cessation clinical trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 108 (Estimated)
Dates: Start 2025-01-29 (Actual); Primary Completion 2031-08-15 (Estimated); Study Completion 2031-09-30 (Estimated)

PRIMARY OUTCOMES:
Focus Groups | Baseline
  Audio recordings will be analyzed by the research team using a template-based rapid analysis technique developed for health services research. A structured summary will be prepared, organized by topical areas drawn from the interview/focus group guide, to identify and describe themes within each topical domain.
Veteran Nicotine and Tobacco Use Questionnaire | Phase 1, Baseline
  Assesses age at first use, duration of use, use of all forms of nicotine and tobacco, prior quit attempts (defined as a period of intentionally not smoking for 24 hours), duration of cessation (if any), and presence of other tobacco users in the home. It will be used in the analytic process to correlate findings/themes with characteristics.
Smoking Knowledge, Attitudes and Practices Scale (S-KAP) | Phase 1, Baseline
  It is a validated 46 item instrument that evaluates smoking-related knowledge, beliefs, self-efficacy, cessation treatment practices, and barriers to cessation treatment delivery among healthcare providers. The scores are from the summed items. Higher scores equal more tobacco treatment and the range of scores is 0-26.
Participant Demographic Questionnaire | Phases 2 & 3, Week 0
  Assesses age, gender identity, sexual orientation, ethnicity, race, relationship status, income, education level, military history, service-connected disability status, housing status, and employment status. It will be analyzed through bivariate associations with outcomes (attendance, rate of video uploads).
Session Attendance | Phases 2 & 3, Up to 5 Weeks
  Study engagement will be assessed by tracking the number of participants attend each intervention session over the course of the 5-week intervention period. It will be analyzed through bivariate associations with participant demographics. Differences over time in measurements will be examined using generalized mixed models.
Remote (mobile) CO monitoring | Phases 2 & 3, Weeks 2-5
  Study engagement will be assessed by the proportion of videos uploaded. Videos will be uploaded from Monday to Friday. It will be analyzed through bivariate associations with participant demographics. Differences over time in measurements will be examined using generalized mixed models.
Recruitment yield number of participants enrolled | Phases 2 & 3, Up to 5 Weeks
  Study feasibility will be assessed by recruitment yield, i.e., tracking the number of participants who initiated treatment.
Study Retention | Phases 2 & 3, 5 weeks
  Study retention as assessed by the number of participants that completed the study.
Timeline Follow-Back (TLFB): TUD medication | Phase 3, Weeks 0, 5, 12, 24
  Self-reported use of medication for tobacco use disorder will be assessed with TLFB, which uses a calendar with specific anchor dates to identify the quantity and frequency of use.
Change in Score on the Contemplation Ladder | Phase 3, Weeks 0, 5, 12, 24
  The Contemplation Ladder is a visual analog comprised of 11 rungs and 5 anchor statements, representing stages of change. The response options (0) to (3) corresponded with the stage of precontemplation, (4) to (6) represented the stage of contemplation, (7) and (8) referred to the stage of preparation, (9) and (10) represented the stage of action and stage of maintenance respectively. It is a brief measure of motivation or readiness to change, where (0) is the least motivated and (10) is the most motivated. This measure has been validated for cigarette and other substance use.
Changes in Nicotine and Tobacco Use Survey | Phase 3, Weeks 0, 5, 12, 24
  Assesses age at first use, duration of use, use of all forms of nicotine and tobacco, prior quit attempts (defined as a period of intentionally not smoking for 24 hours), duration of cessation, and presence of other tobacco users in the home and will be completed in Week 0. At Follow Ups (Weeks 5, 12 and 24), the survey will inquire about frequency and duration of quit attempts
Change in Scores on the Fagerström Test for Nicotine Dependence (FTND) | Phase 3, Weeks 0, 5, 12, 24
  The Fagerström Test for Nicotine Dependence is a standard instrument for assessing the intensity of physical addiction to nicotine. It contains six items that evaluate the quantity of cigarette consumption, the compulsion to use, and dependence. In scoring the Fagerström Test for Nicotine Dependence, yes/no items are scored from 0 to 1 and multiple-choice items are scored from 0 to 3. The items are summed to yield a total score of 0-10. The higher the total Fagerström score, the more intense is the patient's physical dependence on nicotine.
Change in Scores on the Questionnaire on Smoking Urges (QSU-Brief) | Phase 3, Weeks 0, 5, 12, 24
  The QSU-Brief consists of 10 statements about the respondent's feelings and thoughts about his or her desire to smoke cigarettes as he or she is completing the questionnaire (i.e., right now). Each response is scored a number ranging from 1 (strongly disagree) to 7 (strongly agree) and scores are calculated by summing the item scores. The higher the total QSU score, the more intense are the participant's smoking urges.
Change in Timeline Followback (TLFB): Tobacco | Phase 2 Weeks 0-6; Phase 3, Weeks 0-24
  Weekly self-reported use of cigarettes will be assessed with TLFB which uses a calendar with specific anchor dates to identify the quantity and frequency of use.
Change in carbon monoxide (CO) levels | Phases 2- 3, Weeks 2-5
  An iCO CO monitor will be used for the bio-verification of cigarette abstinence. Exhaled CO will be obtained using a study-issued iPad equipped with the iCO CO monitor and compatible app and the results will be shared through videos uploaded using VA-provided apps. Participants that report not smoking in the past 7 days and have CO levels <6 parts per million (ppm) will be considered abstinent. For individuals with CO levels> 6 ppm that report smoking cannabis who are not receiving NRT, salivary cotinine <10 nanograms/ milliliter (ng/ml) will be used.

SECONDARY OUTCOMES:
Timeline Follow-Back (TLFB): Other substances | Phase 2 Weeks 0-6; Phase 3, Weeks 0-24
  Self-reported use of other substances will be assessed with TLFB, which uses a calendar with specific anchor dates to identify the quantity of use.
Change in Timeline Follow-Back (TLFB): TUD medication | Phase 2 Weeks 0-6
  Self-reported use of medication for tobacco use disorder will be assessed with TLFB, which uses a calendar with specific anchor dates to identify the frequency of use.
Change in Timeline Follow-Back (TLFB): E-cigarettes | Phase 2 Weeks 0-6; Phase 3, Weeks 0-24
  Self-reported use of e-cigarettes will be assessed with TLFB, which uses a calendar with specific anchor dates to identify the quantity of use.
Change in Timeline Follow-Back (TLFB): Other tobacco products | Phase 2 Weeks 0-6; Phase 3, Weeks 0-24
  Self-reported use of any other tobacco products will be assessed with TLFB, which uses a calendar with specific anchor dates to identify the quantity of use.
Change in Percentage of Participants with Point Prevalent Abstinence | Phase 2, Week 5; Phase 3, Weeks 5-24
  Seven-day point prevalence cigarette abstinence will be defined as the percentage of participants who have reported no smoking or nicotine use on the 7 consecutive days prior to the assessment with biochemically verified cotinine levels of < 10 nanograms/ milliliter.
Mean Salivary Cotinine Levels | Phase 2 Weeks 2-6; Phase 3 Weeks 2-6, 12, and 24
  Salivary Cotinine levels are an established method to biochemically verify a participant's smoking status. Participants will follow instructions provided to them in plain language describing procedures to test saliva for the presence or absence of cotinine to confirm abstinence. The cotinine test has several zones (0-6). Any result of with color in Zone 0 will be considered negative for tobacco use.

CONTACTS AND LOCATIONS:
Overall Officials: Ellen Herbst, MD, Principal Investigator — San Francisco VA Medical Center, San Francisco, CA
Locations (1):
- San Francisco VA Medical Center, San Francisco, CA, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Provides Link to CM_TUD_Cancer Study — https://addictionresearch.ucsf.edu/